CLINICAL TRIAL: NCT05216302
Title: Prehabilitation Program Based on Health Education and Nordic Walking to Reduce Musculoskeletal Impairments in Women Undergoing Breast Cancer Surgery
Brief Title: Prehabilitation for Breast Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Raquel Sebio (Other)
Collaborators: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor-Investigator, Raquel Sebio, Principal Investigator, Universitat Pompeu Fabra
Organization: Universitat Pompeu Fabra (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IIBSP-PRO-2021-10
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
Keywords: breast cancer; prehabilitation; exercise therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (No Intervention): Patients allocated to this arm will continue with their schedule chemotherapy with no additional intervention
- Prehabilitation (Experimental): Patients allocated to this arm will participate in a weekly group-based exercise intervention (nordic walking) and receive health education through a booklet, videos of the exercises and face-to-face sessions prior to each nordic walking session. Chemotherapy will continue as scheduled.
  Interventions: Behavioral: Group-based Nordic Walking Exercise Program

INTERVENTIONS:
Behavioral: Group-based Nordic Walking Exercise Program — An exercise intervention based on nordic walking and health education of one hour and 15 minutes per session. Each session includes 10 min of health education followed by 15 minutes of warm-up exercises, 30 minutes of nordic walking and finally 15 min to cool-down. The intervention is meant to last during two months (last round of chemotherapy and one month pre-surgery), twice weekly for approximately a total of 16 sessions.
  Arms: Prehabilitation

SUMMARY:
Prehabilitation for women diagnosed with breast cancer is commonly not part of the clinical pathways as little time (usually a few days) is left between diagnosis and surgery. However, a great proportion of these patients will undergo neoadjuvant chemotherapy which provides a window opportunity to improve patients' physical status to withstand surgery and minimize post-operative musculoskeletal complications associated with surgery.

To this end, the aim of this study is to assess the efficacy of a prehabilitation program consisting of health education and a supervised nordic walking-based intervention in women diagnosed with breast cancer currently undergoing neoadjuvant chemotherapy to decrease post-operative musculoskeletal impairments and improve functionality of the affected arm.

The study is an open-label, single-blind randomised controlled trial conducted at one tertiary hospital. Women diagnosed with breast cancer scheduled for surgery and currently undergoing chemotherapy will be randomised to either usual care (UC) or prehabilitation (PREHAB). Patients will be assessed for eligibility during the fourth out of six course of chemotherapy. Those randomised to the PREHAB group will participate in a supervised group-based nordic walking intervention twice weekly during 8 weeks (approximately 16 sessions). In addition, participants will receive written information regarding the benefits of exercise during cancer treatment and surveillance. Patients will be assessed prior to surgery as well as at 1, 3 and 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast cancer scheduled for surgery with or without lymphadenectomy
* Candidates to receive neoadjuvant chemotherapy
* Not currently undergoing any other physical therapy therapies or treatments

Exclusion Criteria:

* Cognitive impairment or inability to read Catalan or Spanish
* Prior diagnosis of shoulder impairment or injury
* Major musculoskeletal, neurological or cardiorespiratory limitations to prevent participation in the exercise program

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Disabilities of the Arm Shoulder and Hand Questionnaire (Quick DASH) | Pre-Surgery (one week)
  Functionality of the affected upper arm using the DASH questionnaire. The questionnaire compromises 11 items. Scoring ranges from 0 (no disability) to 100 (more severe disability)
Disabilities of the Arm Shoulder and Hand Questionnaire (Quick DASH) | One month post-surgery
  Functionality of the affected upper arm using the DASH questionnaire. The questionnaire compromises 11 items. Scoring ranges from 0 (no disability) to 100 (more severe disability)
Disabilities of the Arm Shoulder and Hand Questionnaire (Quick DASH) | Three months post-surgery
  Functionality of the affected upper arm using the DASH questionnaire. The questionnaire compromises 11 items. Scoring ranges from 0 (no disability) to 100 (more severe disability)
Disabilities of the Arm Shoulder and Hand Questionnaire (Quick DASH) | Six months post-surgery
  Functionality of the affected upper arm using the DASH questionnaire. The questionnaire compromises 11 items. Scoring ranges from 0 (no disability) to 100 (more severe disability)

SECONDARY OUTCOMES:
Upper arm volume | Pre-Surgery (one week)
  Perimeter of the affected arm will be measured with a tape measure at hand, wrist, elbow and shoulder level
Upper arm volume | One month post-surgery
  Perimeter of the affected arm will be measured with a tape measure at hand, wrist, elbow and shoulder level
Upper arm volume | Three months post-surgery
  Perimeter of the affected arm will be measured with a tape measure at hand, wrist, elbow and shoulder level
Upper arm volume | Six months post-surgery
  Perimeter of the affected arm will be measured with a tape measure at hand, wrist, elbow and shoulder level
Range of Movement (ROM) | Pre-Surgery (one week)
  Range of movement of the affected arm in three axes using a goniometer
Range of Movement (ROM) | One month post-surgery
  Range of movement of the affected arm in three axes using a goniometer
Range of Movement (ROM) | Three months post-surgery
  Range of movement of the affected arm in three axes using a goniometer
Range of Movement (ROM) | Six months post-surgery
  Range of movement of the affected arm in three axes using a goniometer
Pain severity | Pre-Surgery (one week)
  Global pain assessed with a Visual Analog Scale (0 no pain to 10 maximum pain)
Pain severity | One month post-surgery
  Global pain assessed with a Visual Analog Scale (0 no pain to 10 maximum pain)
Pain severity | Three months post-surgery
  Global pain assessed with a Visual Analog Scale (0 no pain to 10 maximum pain)
Pain severity | Six months post-surgery
  Global pain assessed with a Visual Analog Scale (0 no pain to 10 maximum pain)
Health-Related Quality of Life | Pre-Surgery (one week)
  Health-Related Quality of Life will be assessed with the questionnaire developed by the European Organization for Research and Treatment (EORTC) Quality of Life (QLQ) questionnaire (EORTC QLQ C30). Scores range from 0 to 100 with higher values associated with better overall quality of life
Health-Related Quality of Life | One month post-surgery
  Health-Related Quality of Life will be assessed with the questionnaire developed by the European Organization for Research and Treatment (EORTC) Quality of Life (QLQ) questionnaire (EORTC QLQ C30). Scores range from 0 to 100 with higher values associated with better overall quality of life
Health-Related Quality of Life | Three months post-surgery
  HHealth-Related Quality of Life will be assessed with the questionnaire developed by the European Organization for Research and Treatment (EORTC) Quality of Life (QLQ) questionnaire (EORTC QLQ C30). Scores range from 0 to 100 with higher values associated with better overall quality of life
Health-Related Quality of Life | Six months post-surgery
  Health-Related Quality of Life will be assessed with the questionnaire developed by the European Organization for Research and Treatment (EORTC) Quality of Life (QLQ) questionnaire (EORTC QLQ C30). Scores range from 0 to 100 with higher values associated with better overall quality of life
Handgrip Strength | Pre-Surgery (one week)
  Handgrip strength will be determined using an hydraulic dynamometer (Jamar). Both hands will be assessed and the better result out of three attempts will be used.
Handgrip Strength | One month post-surgery
  Handgrip strength will be determined using an hydraulic dynamometer (Jamar). Both hands will be assessed and the better result out of three attempts will be used.
Handgrip Strength | Three months post-surgery
  Handgrip strength will be determined using an hydraulic dynamometer (Jamar). Both hands will be assessed and the better result out of three attempts will be used.
Handgrip Strength | Six months post-surgery
  Handgrip strength will be determined using an hydraulic dynamometer (Jamar). Both hands will be assessed and the better result out of three attempts will be used.
Functional capacity | Pre-surgery (one week)
  Functional capacity will be measured with the distance covered by the 6-Minute Walk Test.
Functional capacity | One month post-surgery
  Functional capacity will be measured with the distance covered by the 6-Minute Walk Test.
Functional capacity | Three months post-surgery
  Functional capacity will be measured with the distance covered by the 6-Minute Walk Test.
Functional capacity | Six months post-surgery
  Functional capacity will be measured with the distance covered by the 6-Minute Walk Test.
Adherence | Pre-Surgery (one week)
  Adherence to the scheduled sessions will be registered in the Prehab group and will be reported as percentage of attended vs. scheduled.
Physical Activity | Pre-surgery (one week)
  Physical activity levels will be measured using the short form of the International Physical Activity Questionnaire (IPAQ). Estimated METS per week will be calculated based on the available formulas.
Physical Activity | One month post-surgery
  Physical activity levels will be measured using the short form of the International Physical Activity Questionnaire (IPAQ). Estimated METS per week will be calculated based on the available formulas.
Physical Activity | Three months post-surgery
  Physical activity levels will be measured using the short form of the International Physical Activity Questionnaire (IPAQ). Estimated METS per week will be calculated based on the available formulas.
Physical Activity | Six months post-surgery
  Physical activity levels will be measured using the short form of the International Physical Activity Questionnaire (IPAQ). Estimated METS per week will be calculated based on the available formulas.

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Sebio, PhD, Study Director — School of Health Sciences TecnoCampus. University Pompeu Fabra
Locations (1):
- Hospital Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Santa Mina D, Brahmbhatt P, Lopez C, Baima J, Gillis C, Trachtenberg L, Silver JK. The Case for Prehabilitation Prior to Breast Cancer Treatment. PM R. 2017 Sep;9(9S2):S305-S316. doi: 10.1016/j.pmrj.2017.08.402. PMID 28942905
- [Background] McNeely ML, Campbell KL, Rowe BH, Klassen TP, Mackey JR, Courneya KS. Effects of exercise on breast cancer patients and survivors: a systematic review and meta-analysis. CMAJ. 2006 Jul 4;175(1):34-41. doi: 10.1503/cmaj.051073. PMID 16818906
- [Background] Silver JK, Baima J. Cancer prehabilitation: an opportunity to decrease treatment-related morbidity, increase cancer treatment options, and improve physical and psychological health outcomes. Am J Phys Med Rehabil. 2013 Aug;92(8):715-27. doi: 10.1097/PHM.0b013e31829b4afe. PMID 23756434
- [Background] Yang A, Sokolof J, Gulati A. The effect of preoperative exercise on upper extremity recovery following breast cancer surgery: a systematic review. Int J Rehabil Res. 2018 Sep;41(3):189-196. doi: 10.1097/MRR.0000000000000288. PMID 29683834
- [Background] ILokapavani Y, Krishna SR, Madhavi K. nfluence of Pre - Operative Physical Therapy Education and Exercise on Post-operative Shoulder Range of Motion and Functional Activites in Subjects with Modified Radical Mastectomy. Int J Physiother 2014. DOI: 10.15621/ijphy/2014/v1i4/54556